CLINICAL TRIAL: NCT02434978
Title: Doppler-guided Endoscopic Treatment in Peptic Ulcer Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Stig Borbjerg Laursen, MD, PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20130140
Record Dates: First submitted 2014-11-12; First posted 2015-05-06 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Peptic Ulcer Bleeding
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplementary doppler-guided endoscopic therapy (Active Comparator)
  Interventions: Device: Supplementary endoscopy with doppler-guided therapy; Drug: IV. PPI; Other: Endoscopic treatment at primary endoscopy
- control group (Placebo Comparator)
  Interventions: Drug: IV. PPI; Other: Endoscopic treatment at primary endoscopy

INTERVENTIONS:
Device: Supplementary endoscopy with doppler-guided therapy — Patients randomized to supplementary doppler-guided therapy undergo repeat endoscopy with doppler evaluation within 24 hours from the primary endoscopy. At the control endoscopy the ulcer base is examined using a doppler device. If active doppler flow is demonstrated the ulcer is treated with a thermal probe until a control doppler-scan is negative. All patients are observed for rebleeding at a specialized GI-bleeding unit.
  Arms: Supplementary doppler-guided endoscopic therapy
Drug: IV. PPI — All patients receive 80mg of Esomeprazole iv as a bolus followed by 8mg Esomeprazole per hour for 72 hours.
Other: Endoscopic treatment at primary endoscopy — All patients are initially treated with endoscopic therapy using a minimum of two different treatment modalities. The primary endoscopy is performed wihtin 24 hours from time of admission to hospital

SUMMARY:
The present study is a randomized controlled trial (RCT) that examines if the outcome of peptic ulcer bleeding could be improved by use of doppler-guided endoscopic treatment.

DETAILED DESCRIPTION:
This study evaluates if performance of a control endoscopy with doppler-guided endoscopic treatment is associated with an improved outcome in term of lower rate of rebleeding and lower rate of bleeding-related mortality. A potential risk of increased risk of complications (in particular perforation) among patients treated with control endoscopy is also evaluated. Outcomes are prospectively registered based on patient records.

ELIGIBILITY:
Inclusion Criteria:

* Peptic ulcer bleeding from ulcers classified as Forrest I-IIb

Exclusion Criteria:

* Severe comorbidity with a remaining life expectancy below 30 days

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-09 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Rebleeding | 1 week
  Number of participants who develop symptoms of rebleeding combined with a significant drop in systolic blood pressure, or B-haemoglobin, or confirmation of stigmata of bleeding at repeat endoscopy/angiography/surgery.

SECONDARY OUTCOMES:
Bleeding-related mortality | 1 month
  Number of participants who die within 30 days from primary endoscopy because of severe rebleeding.
Complications to endoscopic therapy | 1 month
  Number of participants who develop complications to applied endoscopic therapy.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of gastrointestinal surgery, Aalborg University Hospital, Aalborg
  - Department of gastroenterology, Odense University Hospital, Odense